CLINICAL TRIAL: NCT06823323
Title: The Study on the Efficacy and Safety of Lactobacillus Johnsonii in Combination with CapeOX and Pembrolizumab for the Treatment of MSS/pMMR Metastatic Colorectal Cancer- a Prospective, Multicenter, Double-blind, Randomized Controlled Study.
Brief Title: The Study on the Efficacy and Safety of Lactobacillus Johnsonii in Combination with CapeOX and Pembrolizumab for the Treatment of MSS/pMMR Metastatic Colorectal Cancer.
Acronym: MSSpMMRCapeOX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: First Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-0769
Record Dates: First submitted 2025-01-05; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-12

CONDITIONS: Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — CbsT2 protein, Lactobacillus johnsonii

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CapeOX + Pembrolizumab + Lactobacillus johnsonii Group (Experimental): Participants receive CapeOX + Pembrolizumab + Lactobacillus johnsonii
  Interventions: Dietary Supplement: Lactobacillus johnsonii
- CapeOX + Pembrolizumab + Placebo Group (Placebo Comparator): Participants receive CapeOX + Pembrolizumab + Placebo Group
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus johnsonii — It is previously reported Lactobacillus johnsonii #CGMCC29884 in Cell. Animal studies showed it combined with Clostridium sporogenes to produce indolepropionic acid, modulating CD8+ T cell immune quiescence in the tumor microenvironment and sensitizing immunotherapy in CRC, breast cancer, and melanoma. Mager et al. found Lactobacillus johnsonii enhanced CTLA-4 mAb antitumor effects in CRC mouse models. Studies showed it's a typical probiotic widely distributed in various hosts' guts and has long been applied in food and feed industries. Preclinical studies indicated it improved memory through the gut-brain axis, had anti-inflammatory and antibacterial effects, and regulated metabolic diseases. Randomized trials found it effectively inhibited Helicobacter pylori colonization without obvious adverse reactions, suggesting it's a potentially safe and effective treatment.
  Arms: CapeOX + Pembrolizumab + Lactobacillus johnsonii Group
Other: Placebo — Placebo
  Arms: CapeOX + Pembrolizumab + Placebo Group

SUMMARY:
The goal of this clinical trial is to verify the effectiveness and safety of Lactobacillus johnsonii in combination with CapeOX and Pembrolizumab for the treatment of MSS/pMMR metastatic colorectal cancer (CRC). The main questions it aims to answer are:

① To verify the effectiveness of Lactobacillus johnsonii in the treatment of MSS/pMMR type metastatic colorectal cancer (mCRC) who have failed the standard regimen of chemotherapy;

② To explore the safety of Lactobacillus johnsonii in the treatment of MSS/pMMR type metastatic colorectal cancer (mCRC) who have failed the standard regimen of chemotherapy.

Participants who meet all the inclusion criteria will be enrolled in the study and randomly assigned in a 1:1 ratio to either the CapeOX + Pembrolizumab + placebo group or the CapeOX + Pembrolizumab + Lactobacillus johnsonii group.

ELIGIBILITY:
Inclusion Criteria

* Ages between 18 and 75 years old;

  * Pathologically confirmed MSS or pMMR colorectal adenocarcinoma (PCR method, with 0 or 1 locus unstable; or immunohistochemical method, with expression of MLH1/MSH2/MSH6/PMS2 proteins);

    * Patients who have failed standard first- and second-line treatments (including CapeOX ± targeted therapy, FOLFOX ± targeted therapy, 5-FU/LV ± targeted therapy); ④ Radiological imaging indicates distant metastases throughout the body, considered as unresectable lesions; ⑤ Willingness to comply with the study visit schedule, as well as the prohibitions and restrictions stipulated in this agreement.

Exclusion Criteria

* Use of antibiotics within 4 weeks prior to treatment;

  * Concurrent immunodeficiency diseases (such as HIV or post-transplantation status) or receipt of high-dose systemic corticosteroid therapy or any other form of immunosuppressive therapy within the last 4 weeks;

    * Concurrent malignancies in other organs; ④ Concurrent active autoimmune diseases (i.e., requiring corticosteroids or immunosuppressant medications);

      * Concurrent active infections requiring systemic treatment; ⑥ Concurrent severe systemic diseases, diseases of vital organs such as the heart, lungs, and brain, liver and renal insufficiency, among others;

        * Participation in other drug studies within 3 months prior to treatment or inability of the patient to correctly express their chief complaints and cooperate with this study; ⑧ Any severe or uncontrolled medical condition that, in the investigator's opinion, may increase the risks associated with study participation or study drug administration, impair the subject's ability to receive the protocol-specified treatment, or interfere with the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | from randomization to the occurrence of tumor progression or death from any cause, whichever comes first, up to 24 months.
  Progression-Free Survival (PFS), as per RECIST 1.1 criteria, assessed by blinded independent review, is defined as the time from randomization to the occurrence of tumor progression or death from any cause, whichever comes first, up to 24 months.

SECONDARY OUTCOMES:
Objective Response Rate, ORR | from enrollment to the end of treatment, up to 24 months.
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve either a Complete Response (CR) or a Partial Response (PR), as determined by blinded independent review according to RECIST 1.1 criteria.

IPD SHARING:
Plan to Share IPD: No